CLINICAL TRIAL: NCT00473213
Title: Optimizing IFN Beta - 1B Dose
Acronym: Optims
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Collaborators: Dimensione Ricerca s.r.l. (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IFN1B/99
Record Dates: First submitted 2007-05-11; First posted 2007-05-14 (Estimated); Last update posted 2007-05-14 (Estimated); Status verified 2007-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Interferon; Magnetic Resonance
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon-beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Interferon Beta 1

SUMMARY:
BetaferonR is effective in reducing relapse rate and MRI T2-weighted lesion frequency in MS patients at the dose of 8 MIU on alternate days (THE IFNB MS Study Group, 1993). Relapse rate is reduced by 30-35% (The IFNB MS Study Group, 1993), MRI activity is decreased up to 100% in most cases (Stone et al 1995). In some patients, however, MRI activity still occurs or reappears during treatment (Stone et al 1995). MRI activity has been demonstrated to correlate with relapse occurrence (McFarland et al, 1992; Miller et al, 1996), and in some patients relapses still occur during IFN beta treatment. In other patients relapses may occur in association with the appearance, after 9-18 months of treatment, of anti-IFN beta NAB (The IFNB M S Study Group, 1995).

This protocol hypothesizes that the dose of 12 MIU BetaferonR on alternate days has more pronounced MRI and clinical effects in MS patients than that of 8 MIU. MS patients who do not respond to 8 MIU may take advantage of a higher dose. We, therefore decided to assess MRI effects after increasing the Betaferon dose (12 MIU) in RRMS patients showing a residual MRI activity (at least one new Gd enhancing lesion) during six months of standard Betaferon dose treatment (8 MIU).

DETAILED DESCRIPTION:
Comparing the frequency of new Gd enhancing lesions in a group of patients presenting a residual MRI activity during the last four months of the six month standard dose (8MIU) Betaferon treatment randomized to continue the standard dose or to increase the dose to 12 MIU Betaferon

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained.
2. Age between 18 and 50 years inclusive.
3. Male and female patients.
4. Clinically definite or laboratory supported definite RR MS (Poser et al, 1983) for not less than 2 year.
5. Two clinically documented relapses during the preceding 24 months.
6. No relapse or relapse related neurological deterioration for at least 30 days prior to entry in the study.
7. Patients EDSS score from 1 to 3.5 (probably to be extended to 5.5).
8. MRI activity. At least one enhancing lesion during the baseline MRI run-in study .
9. Women capable of having children must agree to use adequate con-traceptive methods (condoms with spermicides, IUCD, oral contraceptives or other adequate barrier contraception).
10. Caregivers agreement to assist the patient to comply with study requirements, if neces-sary (e.g. study drug administration, visits to center).

Exclusion Criteria:

1. Any form of Multiple Sclerosis other than relapsing-remitting.
2. Any other disease which could better explain the patient's signs and symptoms.
3. Any other disabling condition, which could interfere with the clinical evaluation.
4. Pregnancy or lactation.
5. Medical psychiatric, or other conditions that compromise patient's ability to give informed consent, to comply with the trial protocol, or to complete the study.
6. Alcohol or drug abuse in the 90 days preceding screening visit.
7. Uncontrolled clinically significant heart diseases, i.e., cardiac arrhythmias, uncon-trolled angina pectoris, uncompensated congestive heart failure
8. Clinically significant liver, renal and bone marrow dysfunction as defined by the ran-ges of laboratory evaluations. The following ranges (see table 1) for key laboratory evaluations will be considered as adequate for inclusion:

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 217 (Actual)
Dates: Start 1999-09; Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
the effects of BetaferonR on MRI enhancing lesion frequency are detectable very early.Differently from clinical effects on relapse rate, BetaferonR administration results in an almost immediate reduction of enhancing lesion frequency at MRI. | two year

SECONDARY OUTCOMES:
Monitoring MRI effects (evaluating the number of total active lesions, areas of gadolinium-enhancing, T1 hypointense, and T2 hyperintense lesions)Monitoring clinical effects (relapse frequency and severity, changes in EDSS) | two years

CONTACTS AND LOCATIONS:
Overall Officials: Luca Durelli, Prophessor, Study Chair — Università degli studi di Torino-Clinica Neurologica I , Via Cherasco 15 10100 Torino; Antonio Carolei, M D, Principal Investigator — Ospedale Nuovo San Salvatore-Clinica Neurologica .Località Coppito.67100 L'Aquila; Roberto Cavallo, M.D., Principal Investigator — Ospedale Mafggiore San Giovanni Bosco,Divisione di Neurologia Piazza Donatori del Sangue, 3 10154 Torino; Vittorio Cosi, Prophessor, Principal Investigator — Università degli Studi di Parma .Dipartimento di Scienze Neurologiche.Via Palestro 3 27100 Pavia; Luciano Deotto, M.D., Principal Investigator — Ospedale Civile Maggiore, Divisione Neurologica, Piazzale Stefani1 37134 Verona; Claudio Geda, M.D., Principal Investigator — Ospedale Civile di Chivasso.Divisione di Neurologia10034 Chivasso Torino; Giorgio gIULIANI, M.D, Principal Investigator — Ospedale Generale di Macerata,Servizio di Neurofisiopatologia, Via Santa Lucia 1 62100 Macerata.; Angelo Ghezzi, M.D., Principal Investigator — Ospedale SAntonio Abate Servizio recupero Neurologico. Centro Studi S.M. Via Pastore 4 21013 Gallarate (VA); Roberto Cotrufo, M.D., Principal Investigator — Policlinico II Università degli Studi di Napoli. Dipartimento di Neurologia.Piazza Miraglia 2 80138 Napoli; Luigi Murri, Prophessor, Principal Investigator — Università degli Studi di Pisa Clinica Neurologica, Via Roma 67 56100 Pisa; Domenico Caputo, M.D., Principal Investigator — Istituto Don Carlo Gnocchi Divisione Neurologica Riabilitativa. Via Capecelatro 66 20148 Milano; Enrico Montanari, M.D., Principal Investigator — Ospedale Civile di Fidenza, Divisione di Neurologia Via Borghesi 1, 43036 Fidenza (Pr); Franco Perla, M.D., Principal Investigator — Ospedale S. Croce e Carle Divisione di Neurologia, Via Michele Coppino 26, 12100 Cuneo; Federico Piccoli, Prophessor, Principal Investigator — Università degli Studi di Palermo Istituto di Neuropsichiatria, Via Gaetano della Loggia 90129 Palermo; Alessandra Protti, M.D., Principal Investigator — Ospedale Niguarda Cà Granda Divisione Neurologica, Piazza Benefattori 3, 20100 Milano; Giovanni Meola, Prophessor, Principal Investigator — Ospedale Clinico San Donato Neurologia, Via Morandi 30, 20097 San Donato Milanese; Arturo Reggio, Prophessor, Principal Investigator — Policlinico Universitario Centro Sclerosi Multipla, Via S.Sofia 78, 95185 Catania; MariaRosa Rottoli, M.D., Principal Investigator — Ospedali Riuniti di Bergamo Divisione di Neurologia.Largo Barozzi.124100 Bergamo; Elio Scarpini, M.D, Principal Investigator — Università Degli Studi di Milano Istituto di Clinica Neurologica .Via Francesco Sforza 35 20122 Milano; Andrea Spissu, M.D., Principal Investigator — Azienda Ospedaliera G. Brotzu Divisione di Neurologia. Via G. Peretti 90134 Cagliari; Francesco Teatini, M.D., Principal Investigator — Ospedale Generale di Bolzano Divisione di Neurologia Via Lorenz Bohler 5 39100 Bolzano; Riccardo Urciuoli, M.D-, Principal Investigator — Ospedale Silvestrini Divisione di Neurologia 06156 Loc S Andrea delle Fratte Perugia; Luisa Motti, M.D, Principal Investigator — Centro Sclerosi Multipla Divisione di Neurologia Arcispedale S.Maria Nuova, Viale Risorgimento 57 42100 Reggio Emilia; Ruggero Capra, M.D., Principal Investigator — Centro Regionale Sclerosi Multipla Piazzale Spitali Civili 1 25123 Brescia

REFERENCES:
- [Background] Durelli L, Bongioanni MR, Ferrero B, Oggero A, Marzano A, Rizzetto M. Interferon treatment for multiple sclerosis: autoimmune complications may be lethal. Neurology. 1998 Feb;50(2):570-1. doi: 10.1212/wnl.50.2.570. No abstract available. PMID 9484407
- [Derived] Durelli L, Barbero P, Cucci A, Ferrero B, Ricci A, Contessa G, De Mercanti S, Ripellino P, Lapuma D, Viglietta E, Bergui M, Versino E, Clerico M; OPTIMS Trial NAb Sub-Study Group. Neutralizing antibodies in multiple sclerosis patients treated with 375 micrograms interferon-beta-1b. Expert Opin Biol Ther. 2009 Apr;9(4):387-97. doi: 10.1517/14712590902762781. PMID 19278300